CLINICAL TRIAL: NCT06369480
Title: Prognostic Factors for Survival in Patients With Cholangiocarcinoma
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Hans-Christian Pommergaard, Staff Specialist, Department of Surgery and Transplantation, Hepato - Pancreato - Biliary (HPB) team, Rigshospitalet, University of Copenhagen, Rigshospitalet, Denmark
Other Study IDs: Journal-nr.: R-23057752
Record Dates: First submitted 2024-04-11; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Cholangiocarcinoma
Keywords: Cholangiocarcinoma; Survival; Surgery; Treatment
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Surgical Procedures, Operative; Drug Therapy; Neoadjuvant Therapy; Chemotherapy, Adjuvant; Radiotherapy; Palliative Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cholangiocarcinoma: Patients with diagnosis of Cholangiocarcinoma confirmed by MDT
  Interventions: Procedure: Resection/Ablation of tumor; Procedure: Palliative chemotherapy; Procedure: Neoadjuvant chemotherapy; Procedure: Stereotatic radiotherapy; Procedure: Best supportive care

INTERVENTIONS:
Procedure: Resection/Ablation of tumor — Curative treatment
  Other Names: Surgery
Procedure: Palliative chemotherapy — Chemotherapeutic medications
  Other Names: Chemotherapy
Procedure: Neoadjuvant chemotherapy — Chemotherapeutic medications after surgery
  Other Names: Adjuvant chemotherapy
Procedure: Stereotatic radiotherapy — Radiotherapy
  Other Names: Radiotherapy
Procedure: Best supportive care — Symptomatic treatment, non-curative treatment
  Other Names: Supportive care

SUMMARY:
The objective of this retrospective study is to determine the survival rates of CCA patients based on different therapeutic approaches. Additionally, we aim to investigate the risk factors associated with poor survival within a cohort of patients treated over a seven-year period across four Danish hospitals. We anticipate that our findings could provide additional evidence for clinical decision-making, improve patient outcomes, and contribute to the knowledge in the field.

DETAILED DESCRIPTION:
BACKGROUND

Cholangiocarcinoma (CCA) is a highly aggressive neoplasia and is considered the second most common primary liver cancer (1). Its global mortality has shown an upward trend over the last two decades (2), with a survival rate of less than 5% at 5 years. The poor prognosis is related to late-stage detection since CCA can be asymptomatic in its early stages (3). In Denmark, the estimated cumulative risk of mortality due to CCA was 0.74 for men (ranking 20th in all of Europe) and 0.34 for women (ranking 6th in Europe) (4).

CCA is anatomically classified into three groups: intrahepatic, perihilar, and distal CCA (1,2). Additionally, CCA can be classified as mass-forming, periductal infiltrating, and intraductal based on tumor location, which may be associated with tumor morphology (3). A precise anatomical classification of CCA in each case is essential for accurately assessing potential complications (1).

The diagnosis, staging, and treatment of CCA can be challenging and are typically performed by a multidisciplinary team (MDT) of specialists. MDT meetings are a common practice in cancer care aimed at improving survival. However, it is important to note that there are currently no standardized recommendations for MDT practices in CCA (2). Recently, authors have made efforts to identify areas of improvement and establish standard guidelines for MDT decisions based on the current practices of specialized European teams with expertise in CCA. According to the recommendations of the European Network for the Study of Cholangiocarcinoma, international guidelines should be utilized for MDT decisions. However, preference for national guidelines should be given (2) Nevertheless, at the moment, there are not in Denmark a national guideline to determine the most optimal treatment for CCA patients based on local statistics.

Hence, the objective of this retrospective study was to determine the survival rates of CCA patients based on different therapeutic approaches. Additionally, we aimed to investigate the risk factors associated with poor survival within a cohort of patients treated over a seven-year period across four Danish hospitals. We anticipate that our findings could provide additional evidence for clinical decision-making, improve patient outcomes, and contribute to the knowledge in the field.

AIMS AND HYPOTHESIS

Aim I Determine the survival rates of CCA patients based on various therapeutic approaches following the MDT decision.

Aim II Determine the risk factors associated with unfavorable overall survival in CCA patients.

Hypothesis Advanced age, male gender, poor performance status, non-operability, lack of tumor resectability, and being treated in a hospital where the MDT decision is made all pose as poor survival risk factors for CCA patients. In contrast, we anticipate a better prognosis for patients undergoing curative treatment (surgery) compared to non-surgical treatments. Finally, our hypothesis suggests that chemotherapy provides a better prognosis than no treatment in CCA patients.

KEY DATA SOURCES

Primary data sources Patients will be identified in the Danish Liver-Biliary Cancer Database and data was retrieved retrospectively from medical records in individual centers. The Danish Data Protection Agency (p-2023-14848) has approved the study.

Inclusion criteria Patients' eligibility for this study is contingent on a diagnosis of CCA confirmed by the MDT from Aalborg Universitetshospital, Aarhus Universitetshospital, Odense Universitetshospital, and Rigshospitalet in Denmark from 2013 to 2020.

Exclusion criteria We will exclude from the analysis all records resulting from more than one intervention (on the same patient). Additionally, all patients whose cholangiocarcinoma diagnosis was canceled following the MDT meeting were also excluded, as well those with inconsistent data regarding date of reference to the MDT.

DEFINITION OF PRIMARY OUTCOMES Overall survival will be defined as the period from the initial diagnosis of the disease to the registered date of death, regardless of the cause. The disease diagnosis will be determined from the date of MDT referral, and the date of death will be based on the information provided in the Danish Civil Registration (CPR) number.

STATISTICAL ANALYSIS Patient baseline characteristics were described using the mean and standard deviation (SD) for continuous data and frequency and percentage for categorical data. Differences between treatment plan groups in variables with a normal distribution were analyzed with an ANOVA test. Non-normally distributed data were analyzed with Kruskal-Wallis test and presented as medians and interquartile ranges. Overall survival was calculated from the date of referral to the MDT to the date of death reported in the Danish Civil Registration (CPR) number. Survival analysis was conducted using the Kaplan-Meier estimator with a 95% confidence interval. The analysis of risk factors associated with CCA patients' survival was performed using univariate Cox regression analysis. Significance was considered when the P-value was <0.05. All analyses were conducted using SPSS version 29.0.01.1 (171).

ELIGIBILITY:
Inclusion Criteria:

* Patients' eligibility for this study is contingent on a diagnosis of CCA confirmed by the MDT from Aalborg Universitetshospital, Aarhus Universitetshospital, Odense Universitetshospital, and Rigshospitalet in Denmark from 2013 to 2020.

Exclusion Criteria:

* We will exclude from the analysis all records with more than one interventions. Additionally, all patients whose cholangiocarcinoma diagnosis was canceled following the MDT meeting will be also excluded, as well those with inconsistent data regarding date of reference to the MDT.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients identified in the Danish Liver-Biliary Cancer Database with a confirmed diagnosis of cholangiocarcinoma registered from 2013 to 2020.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Aim I | 6 months
  Determine the survival rates of CCA patients based on various therapeutic approaches following the MDT decision.
Aim II | 6 months
  Determine the risk factors associated with unfavorable overall survival in CCA patients.

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Christian Pommergaard, M.D./Ph.D., Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tawarungruang C, Khuntikeo N, Chamadol N, Laopaiboon V, Thuanman J, Thinkhamrop K, Kelly M, Thinkhamrop B. Survival after surgery among patients with cholangiocarcinoma in Northeast Thailand according to anatomical and morphological classification. BMC Cancer. 2021 May 3;21(1):497. doi: 10.1186/s12885-021-08247-z. PMID 33941120
- [Background] Thuehoj AU, Andersen NC, Worm ES, Hoyer M, Tabaksblat EM, Weber B, Mortensen HR. Clinical outcomes after stereotactic ablative radiotherapy in locally advanced cholangiocarcinoma. Acta Oncol. 2022 Feb;61(2):197-201. doi: 10.1080/0284186X.2021.1995893. Epub 2021 Nov 2. No abstract available. PMID 34726565
- [Background] Cillo U, Fondevila C, Donadon M, Gringeri E, Mocchegiani F, Schlitt HJ, Ijzermans JNM, Vivarelli M, Zieniewicz K, Olde Damink SWM, Groot Koerkamp B. Surgery for cholangiocarcinoma. Liver Int. 2019 May;39 Suppl 1(Suppl Suppl 1):143-155. doi: 10.1111/liv.14089. PMID 30843343
- [Background] Moris D, Palta M, Kim C, Allen PJ, Morse MA, Lidsky ME. Advances in the treatment of intrahepatic cholangiocarcinoma: An overview of the current and future therapeutic landscape for clinicians. CA Cancer J Clin. 2023 Mar;73(2):198-222. doi: 10.3322/caac.21759. Epub 2022 Oct 19. PMID 36260350
- [Background] Li Y, Song Y, Liu S. The new insight of treatment in Cholangiocarcinoma. J Cancer. 2022 Jan 1;13(2):450-464. doi: 10.7150/jca.68264. eCollection 2022. PMID 35069894
- [Background] Ma KW, Cheung TT, Leung B, She BWH, Chok KSH, Chan ACY, Dai WC, Lo CM. Adjuvant chemotherapy improves oncological outcomes of resectable intrahepatic cholangiocarcinoma: A meta-analysis. Medicine (Baltimore). 2019 Feb;98(5):e14013. doi: 10.1097/MD.0000000000014013. PMID 30702559